CLINICAL TRIAL: NCT05376943
Title: The Occurrence of HCC and Possible Differences in Its Course Depending on DAA Treatment
Brief Title: Possible Differences in HCC Course Depending on DAA Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: AKBE/118/2021
Record Dates: First submitted 2021-09-27; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-09

CONDITIONS: Carcinoma, Hepatocellular; Hepatitis C Virus Infection, Response to Therapy of; Drug Effect; Drug Side Effect; Hepatitis C, Chronic; Liver Cirrhosis
Keywords: hepatocellular carcinoma; hepatitis C; direct-acting antiviral agents
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C; Drug-Related Side Effects and Adverse Reactions; Hepatitis C, Chronic; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients diagnosed with HCC after receiving direct acting antiviral HCV treatment: In this group there will be patients with the diagnosis of hepatocellular carcinoma, who underwent direct acting antiviral treatment. We will collect both epidemiological (age, gender, comorbidities, alcohol abuse) and clinical data (serum bilirubin, alanine, aspartate aminotransferase, gammaglutamyltransferase, alkaline phosphatase and alpha-fetoprotein level, Child-Pugh and MELD score, imaging tests, liver biopsy and elastography, if performed). The HCV infection and co-infections will be assessed and also the composition of therapy and the response to treatment will be evaluated.
  Interventions: Drug: Direct Acting Antivirals
- Patients diagnosed with HCC who were not receiving direct acting antiviral HCV treatment: In this group there will be patients with the diagnosis of hepatocellular carcinoma, who were not receiving direct acting antiviral treatment. We will collect both epidemiological (age, gender, comorbidities, alcohol abuse) and clinical data (serum bilirubin, alanine, aspartate aminotransferase, gammaglutamyltransferase, alkaline phosphatase and alpha-fetoprotein level, Child-Pugh and MELD score, imaging tests, liver biopsy and elastography, if performed). The HCV infection and co-infections will also be assessed.

INTERVENTIONS:
Drug: Direct Acting Antivirals — Our observational study will assess the exposure to direct acting antivirals - the specific drugs, dose, duration of the therapy and the effect of the treatment.
  Groups: Patients diagnosed with HCC after receiving direct acting antiviral HCV treatment

SUMMARY:
BACKGROUND It is estimated that around 71 milion people live with chronic hepatitis C virus (HCV) infection. This may lead to the development of liver cirrhosis and hepatocellular carcinoma (HCC). Liver cirrhosis is considered as one of the most common risk factors of hepatocellular carcinoma (HCC). HCC is seventh most common cancer worldwide. The treatment of HCV with direct-acting antivirals (DAAs) has led to the increase of sustained virological response (SVR) rates to more than 90%. It is suggested that the virus eradication reduces, but not eliminates the risk of HCC. This concerns especially patients with liver cirrhosis or previous HCC history. There are reports of early occurrence of HCC after the DAA treatment. Therefore, patients undergoing successful HCV treatment should be monitored for the possibility of hepatoccelular carcinoma occurrence.

AIM OF THE STUDY In this study the investigators aimed to assess the occurrence of HCC after direct acting antiviral HCV treatment and evaluate whether the course of HCC and liver function differ among the population of patients treated with DAAs and those who were not receiving the therapy with DAA.

MATERIAL AND METHODS This is the observative, cohort, retrospective study which will be performed in several clinical centres in Poland. The inclusion criteria are: hepatocellular carcinoma diagnosis, age >18 years old.

The investigators will collect both epidemiological (age, gender, comorbidities, alcohol abuse) and clinical data (serum bilirubin, alanine, aspartate aminotransferase, platelets, gammaglutamyltransferase, alkaline phosphatase and alpha-fetoprotein level, Child-Pugh and MELD score, imaging tests, liver biopsy and elastography, if performed).

In all patients, the HCV infection and co-infections will be assessed. In those who underwent the DAA treatment, the composition of the therapy and response to the treatment will be evaluated.

Statistical analysis will be performed in subgroups of patients undergoing DAA treatment and without the therapy. The distribution of continuous variables will be analysed by the Shapiro-Wilk test. Quantitative data will be analysed using the Mann-Whitney U test or Kruskal-Wallis ANOVA when appropriate. Qualitative data will be compared using the χ² test or the Fisher exact test. Correlations between quantitative variables will be assessed using the Spearman correlation coefficient. P value will be set at <0.05.

FUNDING:

No remuneration is provided for participation in the study

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma diagnosis
* age >18 years old

Exclusion Criteria:

* age <18 years old

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected from several clinical centres in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The occurrence of HCC after direct acting antiviral HCV treatment. | 1 year

SECONDARY OUTCOMES:
The comparison of the course of HCC among the population of patients treated with DAAs and those who were not receiving the therapy. | 1 year
The difference in liver function tests among the population of patients treated with DAAs and those who were not receiving the therapy. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland